CLINICAL TRIAL: NCT01049646
Title: Interaction of Apelin and Angiotensin in the Systemic Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Dr Gareth Barnes, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FS/09/019/26905 - 2
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Renin Angiotensin System
Keywords: renin-angiotensin system; apelin; systemic haemodynamics
MeSH Terms: interventions — Angiotensin II; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angiotensin II (Active Comparator)
  Interventions: Drug: Angiotensin II
- Saline infusion (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Angiotensin II — Infusion of a subpressor dose of angiotensin II will be give, this will be 0.5microG/min/kg. Thereafter thre ascending doses of apelin will be given, during which time cardiac output and systemic haemodynamics will be measured.
  Arms: Angiotensin II
Drug: Saline — Infusion of saline. Thereafter three ascending doses of apelin will be given, during which time cardiac output and systemic haemodynamics will be measured.
  Arms: Saline infusion

SUMMARY:
The apelin-APJ system is a relatively new discovery. It has generated interest in part due to it's apparent ability to counteract the renin-angiotensin system, which is frequently overactive in many cardiovascular disease.

Apelin improves that pumping ability of the heart and we wish to know if this action persists in the presence of increased levels of angiotensin II.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Healthy volunteers

Exclusion Criteria:

* Lack of informed consent
* Age < 18 years,
* Current involvement in other research studies,
* Systolic blood pressure >190 mmHg or <100 mmHg
* Malignant arrhythmias
* Renal or hepatic failure
* Haemodynamically significant aortic stenosis
* Severe or significant co morbidity
* Women of childbearing potential.

Any regular medication

* Previous history of any cardiovascular disease

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Cardiac output | 90 mins

SECONDARY OUTCOMES:
Systemic haemodynamics | 90mins

CONTACTS AND LOCATIONS:
Locations (1):
- Clincial Research Facility, Royal Infirmary of Edinburgh, 51 Little France Cresc, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Barnes GD, Alam S, Carter G, Pedersen CM, Lee KM, Hubbard TJ, Veitch S, Jeong H, White A, Cruden NL, Huson L, Japp AG, Newby DE. Sustained cardiovascular actions of APJ agonism during renin-angiotensin system activation and in patients with heart failure. Circ Heart Fail. 2013 May;6(3):482-91. doi: 10.1161/CIRCHEARTFAILURE.111.000077. Epub 2013 Mar 21. PMID 23519586